CLINICAL TRIAL: NCT03919747
Title: The Awareness About Oral Contraceptives in Reproductive Age Women
Brief Title: Oral Contraceptives in Reproductive Age Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Mine Kiseli, Assoc. Prof., Ufuk University
Other Study IDs: 20180528/4
Record Dates: First submitted 2019-03-16; First posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Contraception Behavior
Keywords: oral contraceptives; knowledge
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Contraception is an important issue in public health; especially when maternal risks and morbidities are considered. There is a need for consciousness about the contraceptive choices. The reproductive age women in Turkey may be stubborn or may choose to believe heath information. The oral contraceptive drugs are not used because of wrong beliefs. This survey study aims to investigate the consciousness and knowledge about the oral contraceptives in 3 different areas in Turkey.

DETAILED DESCRIPTION:
In this study; surveys will be given to reproductive age women admitting to the obstetrics and gynecology departments in 3 different cities of Turkey. Survey questions start with the education and socioeconomical status of the participants. Mainly the questions include the knowledge, ever use about oral contraceptives.

ELIGIBILITY:
Inclusion Criteria: The women admitting to the clinics -

Exclusion Criteria:

-

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women are the investigation group
Study Population: Reproductive aged women
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-06-02 (Estimated); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge about oral contraceptives | 6 months of survey study
  The number of participants who had knowledge about the correct use of OC pills
Contraindications of OC pills | 6 months of survey study
  The number of participants who know the contraindications of OC pills /The number of participants who think that OC pills cause infertility

SECONDARY OUTCOMES:
Knowledge difference in between different regions | 6 months of survey study
  The number of participants who had knowledge about the correct use of OC pills in different regions
Oral contraceptive use | 6 months of survey study
  The number of participants that have ever used oral contraceptive pills

CONTACTS AND LOCATIONS:
Overall Officials: Recai Pabuccu, Prof., Study Director — The Turkish Reproductive Medicine Association
Locations (3):
- Turkey (Türkiye) (3):
  - Karabuk University Hospital, Karabük
  - Acıbadem Private Hospital, Kayseri
  - Ufuk University Dr Ridvan Ege Hospital, Ankara, Çankaya